CLINICAL TRIAL: NCT04690387
Title: Adaptive Phase I Clinical Trial of Preventive Vaccine Consisting of Autologous Dendritic Cells Previously Incubated With S-protein From SARS-CoV-2, in Subjects Negative for COVID-19 Infection and Anti-SARS-CoV-2 Antibodies
Brief Title: Dendritic Cell Vaccine, AV-COVID-19, to Prevent COVID-19 Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aivita Biomedical, Inc. (Industry)
Collaborators: PT AIVITA Biomedika Indonesia (Unknown); Indonesia Ministry of Health (Unknown); National Institute of Health Research and Development, Ministry of Health Republic of Indonesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CL-COV-P01-ID
Record Dates: First submitted 2020-12-28; First posted 2020-12-30 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — AV-COVID-19 vaccine; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- 0.1 mg antigen, 0 mcg GM-CSF (Experimental): Dendritic cells previously incubated with 0.1 mcg antigen
  Interventions: Biological: AV-COVID-19
- 0.33 mg antigen, 0 mcg GM-CSF (Experimental): Dendritic cells previously incubated with 0.33 mcg antigen
  Interventions: Biological: AV-COVID-19
- 1.0 mg antigen, 0 mcg GM-CSF (Experimental): Dendritic cells previously incubated with 1.0 mcg antigen
  Interventions: Biological: AV-COVID-19
- 0.1 mg antigen, 250 mcg GM-CSF (Experimental): Dendritic cells previously incubated with 0.1 mcg antigen, admixed with 250 mcg GM-CSF
  Interventions: Biological: AV-COVID-19; Other: GM-CSF
- 0.33 mg antigen, 250 mcg GM-CSF (Experimental): Dendritic cells previously incubated with 0.33 mcg antigen, admixed with 250 mcg GM-CSF
  Interventions: Biological: AV-COVID-19; Other: GM-CSF
- 1.0 mg antigen, 250 mcg GM-CSF (Experimental): Dendritic cells previously incubated with 1.0 mcg antigen, admixed with 250 mcg GM-CSF
  Interventions: Biological: AV-COVID-19; Other: GM-CSF
- 0.1 mg antigen, 500 mcg GM-CSF (Experimental): Dendritic cells previously incubated with 0.1 mcg antigen, admixed with 500 mcg GM-CSF
  Interventions: Biological: AV-COVID-19; Other: GM-CSF
- 0.33 mg antigen, 500 mcg GM-CSF (Experimental): Dendritic cells previously incubated with 0.33 mcg antigen, admixed with 500 mcg GM-CSF
  Interventions: Biological: AV-COVID-19; Other: GM-CSF
- 1.0 mg antigen, 500 mcg GM-CSF (Experimental): Dendritic cells previously incubated with 1.0 mcg antigen, admixed with 500 mcg GM-CSF
  Interventions: Biological: AV-COVID-19; Other: GM-CSF

INTERVENTIONS:
Biological: AV-COVID-19 — Autologous dendritic cells previously incubated with SARS-CoV-2 spike protein
Other: GM-CSF — GM-CSF as an adjuvant
  Arms: 0.1 mg antigen, 250 mcg GM-CSF; 0.1 mg antigen, 500 mcg GM-CSF; 0.33 mg antigen, 250 mcg GM-CSF; 0.33 mg antigen, 500 mcg GM-CSF; 1.0 mg antigen, 250 mcg GM-CSF; 1.0 mg antigen, 500 mcg GM-CSF

SUMMARY:
This is an adaptive Phase I trial of a vaccine consisting of autologous dendritic cells previously loaded ex vivo with SARS-CoV-2 spike protein, with or without GM-CSF, to prevent COVID-19 in adults.

DETAILED DESCRIPTION:
Subjects eligible for treatment will be those who at baseline, are not actively infected with SARS-CoV-2, have no evidence of prior infection with SARS-CoV- 2 based on serologic testing, and give informed consent for a vaccination with AV-COVID-19. The patient population will include the elderly and others at higher risk for poor outcomes after COVID-19 infection. For this reason, individuals will not be excluded solely on the basis of age, body mass index, history of hypertension, diabetes, cancer, or autoimmune disease.

After enrolling for screening, subjects will undergo a nasal swab test to exclude active COVID-19 infection and a rapid test for anti-coronavirus antibodies to exclude pre-existing anti-SARS-CoV-2 antibodies. 50 mL of blood will be collected, from which peripheral blood monocytes will be isolated and differentiated into DC before incubation with SARS-CoV-2 S-protein, during which time the protein is digested into 9 to 25 amino acid peptide sequences presented on the dendrites of DC in conjunction with histocompatibility class I and class II molecules. Safety and quality testing will be performed on a small quantity of the batch, and the remaining AV-COVID-19 will be cryopreserved for shipping to the treatment site.

Once the Study Drug is ready, if eligible, the subject will be seen at Study Week-0 for treatment. Prior to injection of the Study Drug, a nasal swab test will be collected to confirm that they are still negative for COVID-19, and blood will be drawn to determine baseline levels of anti-SARS-CoV-2 antibodies. At the treatment site, the product will be thawed and admixed with saline or (saline with GM-CSF), and within 5 hours of thawing, will be injected SC via a 25- gauge needle

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, relatively good health, negative for pre-existing SARS-CoV-2 antibodies, negative for SARS-CoV-2 infection

Exclusion Criteria:

* Active COVID-19 infection by PCR testing, pre-existing SARS-CoV-2 antibodies, pregnant, known hypersensitivity to GM-CSF, known immune deficiency disease, on active treatment with immunosuppressive agent or corticosteroid, participated in previous COVID-19 trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (safety) | 1 week
  Collection of adverse event incidence and severity in all treatment arms

SECONDARY OUTCOMES:
Establish optimal dose formulation | 1 month
  Measurement of antibodies in subject blood
Duration of detection of antibodies against SARS-CoV-2 | 1 month
  Measurement of antibodies in subject blood

CONTACTS AND LOCATIONS:
Overall Officials: Robert O Dillman, MD, Study Chair — Aivita Biomedical, Inc.
Locations (1):
- Rumah Sakit Umum Pusat Dr. Kariadi, Semarang, Central Java, Indonesia